CLINICAL TRIAL: NCT06674980
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Assessing the Efficacy of Human Placental Membrane Products and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers and Venous Leg Ulcers.
Brief Title: Clinical Trial Assessing Human Placental Membrane Products and Standard of Care Versus Standard of Care in Nonhealing DFUs and VLUs
Acronym: C5CAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C5 Biomedical (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00082457
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pathologic Processes; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Disease; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases; Leg Ulcer; Skin Ulcer; Skin Diseases; Diabetes Complications; Diabetic Neuropathies; Foot Diseases; Diabetic Foot; Foot Ulcer; Diabetes Mellitus, Type 2; Ulcer; Foot Ulcer Unhealed
Keywords: Human Placental Membrane (HPM); Diabetic Foot Ulcer (DFU); Venous Leg Ulcer (VLU); Cellular, Acellular, and Matrix-like Product (CAMP); Cellular and/or Tissue-Based Product (CTP)
MeSH Terms: conditions — Pathologic Processes; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetic Angiopathies; Vascular Diseases; Cardiovascular Diseases; Leg Ulcer; Skin Ulcer; Skin Diseases; Diabetes Complications; Diabetic Neuropathies; Foot Diseases; Diabetic Foot; Foot Ulcer; Diabetes Mellitus, Type 2; Ulcer; Varicose Ulcer

STUDY DESIGN:
Masking Description: In addition to the principal investigator's determination of complete closure an independent assessment of the primary endpoint will be performed. Two wound care specialists not associated with the trial ("The Reviewers") will review the digital images of ulcers that have healed. They will review the closed visit and the closure confirmation visit. Deidentified digital images taken with the imaging device will be provided to the reviewers. Two reviewers will assess each photograph and be blinded to the arm in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standard of Care - DFU (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings. Off-loading using the off-loading boot or total contact cast (TCC).
  Interventions: Other: Standard of Care - DFU
- AM/Single - DFU (Experimental): AM/Single is an air-dried, sterile single layer human amniotic membrane allograft.
  Interventions: Other: AM/Single - DFU
- AM/Double - DFU (Experimental): AM/Double is an air-dried, sterile double layer human amniotic membrane allograft.
  Interventions: Other: AM/Double - DFU
- Standard of Care - VLU (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings. Compression using multilayer compression wraps.
  Interventions: Other: Standard of Care - VLU
- AM/Single - VLU (Experimental): AM/Single is an air-dried, sterile single layer human amniotic membrane allograft.
  Interventions: Other: AM/Single - VLU
- AM/Double - VLU (Experimental): AM/Double is an air-dried, sterile double layer human amniotic membrane allograft.
  Interventions: Other: AM/Double - VLU

INTERVENTIONS:
Other: Standard of Care - DFU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care - DFU
Other: AM/Single - DFU — Participants will receive weekly applications of AM/Single and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: AM/Single - DFU
Other: AM/Double - DFU — Participants will receive weekly applications of AM/Double and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: AM/Double - DFU
Other: Standard of Care - VLU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and compression) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: Standard of Care - VLU
Other: AM/Single - VLU — Participants will receive weekly applications of AM/Single and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: AM/Single - VLU
Other: AM/Double - VLU — Participants will receive weekly applications of AM/Double and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: AM/Double - VLU

SUMMARY:
The purpose of the study is to evaluate the efficacy of multiple human placental membrane products and Standard of Care (SOC) versus SOC alone in the management of nonhealing diabetic foot ulcers (DFUs) and venous leg ulcers (VLUs) over 12 weeks using a modified platform trial design.

DETAILED DESCRIPTION:
The C5CAMP trial is a multicenter, prospective, randomized controlled clinical trial to evaluate subjects that meet medical necessity criteria for cellular, acellular, and matrix-like products (CAMPs). The study utilizes a prospective modified platform design to evaluate two separate CAMPs, AM/Single and AM/Double in a single trial. The initial plan is to evaluate two CAMPs; however, the modified platform design permits the inclusion of additional CAMPs. This study will evaluate the clinical utility of multiple CAMPs in the closure of diabetic foot ulcers and venous leg ulcers in subjects in comparison to Standard of Care treatment.

ELIGIBILITY:
Inclusion Criteria for DFU:

1. At least 18 years of age or older.
2. Must have diagnosis of type 1 or 2 Diabetes mellitus.
3. At enrollment, subject must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 20.0 cm2 measured post debridement with the imaging device.
4. Must have a target ulcer that has been present for a minimum of 4 weeks and maximum of 52 weeks of standard of care, prior to screening visit.
5. Target ulcer located on the foot with at least 50% of the ulcer below the malleolus.
6. Target ulcer that is Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
7. Subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and <= 1.3
   2. TBI >= 0.6
   3. TCOM >= 40 mmHg
   4. PVR: biphasic
8. If subject has two or more ulcers, they must be separated by 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcer must be located on the plantar aspect of the foot and must be offloaded for at least 14 days prior to enrollment.
10. Subject must consent to using the prescribed offloading method for the duration of the study.
11. Subject must agree to attend weekly study visits.
12. Subject must be willing and able to participate in the consent process.

Exclusion Criteria for DFU:

1. Subject is known to have a life expectancy of < 6 months.
2. Subject's target ulcer is not secondary to diabetes.
3. Target ulcer is infected or there is cellulitis in the surrounding skin.
4. Target ulcer exposes tendon or bone.
5. Evidence of osteomyelitis complicating the target ulcer.
6. Infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
7. The subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
8. Subject is taking hydroxyurea.
9. Subject has applied topical steroids to the ulcer surface within one month of initial screening.
10. Subject has a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
11. Subject has a glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
12. The surface area of the subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
13. The surface area measurement of the subject's target ulcer decreases by 20% or more during the active 2-week screening phase.
14. Subject has acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
15. Subject is a woman who is pregnant or considering becoming pregnant in the next 6 months.
16. Subject has end stage renal disease requiring dialysis.
17. Subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
18. The subject, in opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
19. Subject was treated with hyperbaric oxygen therapy or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to screening.
20. Subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.

Inclusion Criteria for VLU:

Potential subjects are required to meet all the following criteria for enrollment in the study.

1. Subjects must be at least 18 years of age or older.
2. At randomization subjects must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 20 cm2 measured post-debridement.
3. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
4. No visible signs of healing objectively, less than 40% reduction in wound size in the last 4 weeks.
5. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
6. If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
7. The potential subject must agree to attend the weekly study visits required by the protocol.
8. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria for VLU:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
3. The target ulcer exposes tendon or bone.
4. There is evidence of osteomyelitis complicating the target ulcer.
5. The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
6. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
7. The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
8. The surface area of the target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit ("historical" run-in period). Imaging Device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable).
9. The surface area measurement of the target ulcer decreases by 20% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV-1) to the TV-1 visit during which time the potential subject received SOC.
10. Women who are pregnant or considering becoming pregnant within the next 6 months.
11. The potential subject has end stage renal disease requiring dialysis.
12. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
13. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
14. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
15. The subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
16. A subject has a wound with active or latent infection is excluded.
17. A subject with a disorder that would create unacceptable risk of post-operative complications is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-11-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Determine the percentage of subjects achieving complete closure of target ulcer over 12 weeks. | 1-12 weeks
  The proportion of subjects achieving complete wound closure of target ulcer.

SECONDARY OUTCOMES:
Time to closure for target ulcer. | 1-12 weeks
  Length of time in days to closure will be determined for each treatment group and compared to SOC alone.
Percent Area Reduction (PAR) | 1-12 weeks
  Percent Area Reduction (PAR) will be calculated from Treatment Visit (TV)-1 to TV-13 measured weekly with digital photographic planimetry, using imaging device, and physical examination.
Adverse Events | 1-12 weeks
  Determine number of adverse events
Change in pain in target ulcer | 1-12 weeks
  Change in pain in target ulcer assessed using the Pain, Enjoyment of Life and General Activity (PEG) scale
Determine improvement in quality of life | 1-12 weeks
  Quality of life assessed using the Wound Quality of Life (wQOL) at TV-1, TV-4, TV-8, TV-12 / Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- Poirot Podiatry, Metairie, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No